CLINICAL TRIAL: NCT03917927
Title: A Prospective Multicenter Study of the Integration Success of the Eztetic Dental Implant System in Immediate Loading Cases
Brief Title: A Clinical Study of the Eztetic Dental Implant System
Acronym: RoseQuartz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1601
Record Dates: First submitted 2019-04-13; First posted 2019-04-17 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Eztetic dental implant (Experimental): Eztetic 3.1mm diameter, lengths 8, 10, 11.5, 13, 16 mm
  Interventions: Device: Eztetic dental implant

INTERVENTIONS:
Device: Eztetic dental implant — narrow diameter dental implant

SUMMARY:
This will be a prospective, observational multicenter study. All implants will be placed in the anterior maxilla or mandible and immediately loaded with a provisional prosthesis out of occlusion. Final restorations insertion will take place no later than 6 months following implant placement surgery. All implants will be restored with a single crown or splinted to a pre-existing implant if in the pre-molar region (no 2 adjacent edentulous sites).

DETAILED DESCRIPTION:
This will be a prospective, observational study in which patients in need of dental implants in the anterior regions of the maxilla or mandible will be treated with the Eztetic dental implant(s). Qualified patients will be those with one or more edentulous area in the anterior maxilla or mandible needing a single (restored as a single crown; if in the pre-molar region, it is recommended implant be splinted to another tooth or implant; no 2 adjacent edentulous sites). Qualified patients should have presence of posterior teeth or a stable posterior occlusion. All implants will be placed in a single-stage manner. A provisional abutment will be placed and a temporary crown will be placed (cemented or screw-retained) out of occlusion at implant placement surgery visit. Impressions for permanent prosthesis fabrication will take place at 6 weeks and prosthesis placement will take place at 2 months. Final prosthesis insertion will take place no later than 6 months following implant placement surgery. Resonance frequency assessment procedures will be done at implant placement surgery and at prosthesis insertion. Implant survival will be the primary study endpoint. Crestal bone regression will be the secondary study endpoint. Enrollment will continue until 20 patients have completed final prosthetic treatment at study center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex and at least 18 years of age
2. Patients for whom a decision has already been made to use a dental implant for the restoration of existing partial edentulism in the anterior (central and lateral incisors), canine or pre-molar regions in the mandible or maxilla. Placing implant in canine region should be in a healed site (not for immediate extraction)
3. Immediate extraction or a prior extracted site
4. Intact buccal table as verified by Cone Beam Computed Tomography (CBCT) or radiography during surgery. If absent, patient should be excluded from enrollment in the study.
5. Patients must be physically able to tolerate conventional surgical and restorative procedures.
6. Patients with a facial lingual width of at least 5.1mm and inner tooth width of at least 6mm.
7. Patients having a thick gingival biotype (based on the lack of transparency of the periodontal probe through the gingival margin while probing the buccal sulcus) will be preferred but lack of this characteristic will not disqualify a patient from inclusion in this study.
8. Presence of opposing dentition with a functional occlusion that permits the restoration with a non-occluding provisional prosthesis.
9. Patients who provide a signed informed consent; a patient having implant placement surgery will continue participation in the study regardless of whether or not they receive restorative treatment according to protocol (protocol deviation)
10. Patients who agree to be evaluated for each study visit.
11. Minimum primary stability, insertion torque > 35Ncm (this will be a criteria that is met at the time of surgery)

Exclusion Criteria:

1. Patients with known systemic diseases such as uncontrolled diabetes, endocrine disease, heart disease, immuno-compromised, or mental disorders.
2. Patients with current use of non-steroidal anti-inflammatory drugs, bisphosphonates or corticosteroid treatments.
3. Patients with active infection or severe inflammation in the areas intended for implant placement.
4. Prisoners
5. Patients with a > 10 cigarette per day smoking habit.
6. Patients with a history of therapeutic radiation to the head or jaw.
7. Patients in need of bone grafting at the site of the intended implantation site(s).
8. Patients who are known to be pregnant at the screening visit or planning to become pregnant within 6 months of study enrollment.
9. Patients with evidence of severe parafunctional habits such as bruxing or clenching.
10. Patients with HIV or Hepatitis infection
11. Patients who have previously failed implants at the site intended for study implant placement
12. Patients in need of other treatments or surgeries at a site adjacent to the intended implantation site
13. Patients with a history of severe periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Implant survival | 2 years
  survival (no declaration of failure) of dental implant

SECONDARY OUTCOMES:
Marginal bone changes | 2 years
  Change in bone levels around dental implant

CONTACTS AND LOCATIONS:
Overall Officials: Burak Yilmaz, DDS, Principal Investigator — Ohio State University
Locations (4):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
- San Jose Hospital, Santiago, Chile
- Dr. Tasso-Eyke von Haussen, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No